CLINICAL TRIAL: NCT07297082
Title: Regional Anesthesia in Ambulatory Endovenous Ablation Surgery: Comparison of Postoperative Effects of Femoral Block and Low-Dose Spinal Anesthesia
Brief Title: Regional Anesthesia in Ambulatory Endovenous Ablation Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, İbrahim Topcu, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-266
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Discharge Time; Spinal Anesthesia; Ambulatory Surgery; Femoral Nerve Block
Keywords: Ambulatory surgery; Endovenous laser ablation; Discharge Time; Femoral nerve block; Spinal Anesthesia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Nerve Block (Active Comparator)
  Interventions: Procedure: Femoral nerve block
- Spinal anesthesia (Active Comparator)
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: Femoral nerve block — After monitoring, the patient is in the supine position and the femoral area on the side to be treated is sterilized. A femoral nerve block is then performed using 20 cc of 1% lidocaine using an ultrasound-guided blocking needle.
  Arms: Femoral Nerve Block
Procedure: Spinal anesthesia — After monitoring, patients will be placed in the lateral decubitus position. Following appropriate field sterilization, patients will receive unilateral spinal anesthesia with 6 mg bupivacaine. Five minutes after spinal anesthesia, patients will be placed in the supine position.
  Arms: Spinal anesthesia

SUMMARY:
Varicose veins represent irreversible, abnormal dilatations of the venous structures. They manifest as tortuous, swollen vessels visible beneath the skin of the lower extremities, particularly the feet and legs. Symptoms typically worsen with prolonged standing or sitting. In the early stages, conservative management options-such as the use of compression (elastic) stockings and frequent elevation of the legs-may be effective. In more advanced cases involving extensive varicosities, invasive interventions including sclerotherapy or endovascular ablation may be indicated. These procedures can be performed under local, regional, or general anesthesia.

Spinal anesthesia is a neuraxial technique that produces temporary sensory, motor, and sympathetic blockade through the subarachnoid administration of local anesthetics, with or without adjuvant agents. Clinically, it is commonly employed for surgeries involving the lower extremities, lower abdomen, perineal, gluteal, inguinal, and rectal regions, as well as select urologic and obstetric procedures.

A femoral nerve block is a regional anesthesia technique that involves ultrasound-guided injection of local anesthetic around the femoral nerve in the inguinal region. It provides effective analgesia for the anterior thigh, knee joint, and medial aspect of the lower leg. In endovenous laser ablation (EVLA), a femoral block can offer adequate sensory blockade to serve as a sole anesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score III and above
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Discharge time | On the operation day
  The time (minutes) from the application of spinal anesthesia or femoral nerve block to the patients' discharge will be recorded as the discharge period

SECONDARY OUTCOMES:
Motor block disappearing time | On the operation day
  Time (minutes) to disappearance of complete motor block in the lower extremity
Sensorial block disappearing time | On the operation day
  Time (minutes) to disappearance of sensorial block in the lower extremity

CONTACTS AND LOCATIONS:
Locations (1):
- İbrahim Topcu, Etimesgut, Ankara, Turkey (Türkiye)